CLINICAL TRIAL: NCT00687583
Title: Effect of Head Movement on the Position of Different Tracheal Tubes Determined Radiologically
Brief Title: Head Movement Effect on Different Tracheal Tubes
Status: Withdrawn | Type: Observational
Why Stopped: Research question deemed not of enough clinical importance to proceed.
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Cengiz Karsli, Staff Anesthesiologist, The Hospital for Sick Children
Other Study IDs: 1000010579
Record Dates: First submitted 2008-05-28; First posted 2008-06-02 (Estimated); Last update posted 2016-05-04 (Estimated); Status verified 2016-05

CONDITIONS: Head Movements; Intubation, Intratracheal
Keywords: pediatrics; anesthesia; head movements; endotracheal tube

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
A breathing tube, which is used to secure the airway and allow ventilation of the lungs during general anaesthesia, is inserted into the windpipe either through the nose or mouth. In children, different formulas exist to determine the appropriate size of the tube according to age, and how far it should be advanced into the airway. Head movement can alter the position of the breathing tube, making it go in or come out too far. Different types of breathing tubes may also differ in their change of position with head movement. The aim of this study is to assess the accuracy of the formulae commonly used in our institution for depth of breathing tube placement, and to measure the degree of tube displacement on head movement with different types of tubes.

DETAILED DESCRIPTION:
An endotracheal tube, which is used to secure the airway and allow ventilation of the lungs during general anesthesia, is inserted into the trachea either through the nose or mouth. In children, different formulae exist to determine the approximate size of the tube according to age, and how far it should be advanced into the airway. Once a tracheal tube is inserted, its position is routinely checked to make sure both lungs are ventilated. To prevent displacement, the tube is taped to the lip, chin or at the nose. However, head movement could cause alteration of the tube position, and risk selective endobronchial intubation or inadvertent extubation. Knowledge of how the different tracheal tubes move with head position can help determine the best tube selection to reduce the risk of accidental tube advancement or removal, in cases where certain head positions are required for surgical access.

The aim of this study is to assess the accuracy of the formulae commonly used in our institution for depth of breathing tube placement, and to measure the degree of tube displacement on head movement with different types of tube. Testing the formulae will enable us to be more aware of how frequently inaccurate tube placement may occur. Knowledge of how the different breathing tubes move with head position can help determine the best tube selection to reduce the risk of the tube going in too far or coming out accidentally, for cases were certain head positions are required for surgery.

ELIGIBILITY:
Inclusion Criteria:

* Children undergoing any procedure in the Image Guided Therapy (IGT) department requiring tracheal intubation and chest x-ray

Exclusion Criteria:

* Premature neonates
* Patients with cranio-facial anomalies
* Cervical spine/upper thoracic anomalies
* Laryngomalacia/tracheomalacia
* Chronic hypoxemia (i.e. cardiac conditions with right to left shunts)
* Patients requiring positions other than supine

Ages: 1 Day to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Fifty children undergoing any procedure in the Image Guided Therapy (IGT) department requiring tracheal intubation and chest X-ray, will be recruited and will be evenly distributed in three different age groups (0 to 6 months, 6 to 24 months, 24 months to 6 years).
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2007-04; Primary Completion 2008-12 (Estimated); Study Completion 2009-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Cengiz Karsli, MD, Principal Investigator — The Hospital for Sick Children, Toronto Canada
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada